CLINICAL TRIAL: NCT05750602
Title: Effect of the Food Supplement LIMICOL on LDL Cholesterol and Muscle Function in Subjects Who Undergo a Program of Physical Training (Double-blind, Randomized, Placebo-controlled Study).
Brief Title: Combined Effect of LIMICOL and Physical Activity on LDL Cholesterol and Muscle Function.
Acronym: L2012-12
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lescuyer Laboratory (Industry)
Collaborators: Hopital Gabriel Montpied (Other); Centre de Recherche en Nutrition Humaine d'Auvergne (Other Government); Clinique Médicale Cardio-Pneumologie de Durtol (Unknown); Université d'Auvergne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2013-A00061-44
Record Dates: First submitted 2014-09-08; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Hypercholesterolemia
Keywords: Hypercholesterolemia; LDL cholesterol
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LIMICOL (Experimental): LIMICOL : red yeast rice (with monacolin K, 2 mg), artichoke leaf extract, policosanols, French maritime Pine bark extract, Garlic extract, vitamins E, B2 and B3.
  1 tablet during the 3 principal meals for 12 weeks.
  Interventions: Dietary Supplement: LIMICOL
- PLACEBO (Placebo Comparator): dicalcium phosphate, calcium citrate, vegetable magnesium stearate, microcrystalline cellulose, Maltodextrin, Tricalcium phosphate, Beet powder, Yellow coloring shellac, Brown coloring shellac.
  1 tablet during the 3 principal meals for 12 weeks.
  Interventions: Dietary Supplement: PLACEBO

INTERVENTIONS:
Dietary Supplement: LIMICOL — Suplementation with LIMICOL, 3 tablets per day, together with supervised physical activity (3 times per week) for 12 weeks.
  Arms: LIMICOL
Dietary Supplement: PLACEBO — Suplementation with PLACEBO, 3 tablets per day, together with supervised physical activity (3 times per week) for 12 weeks.
  Arms: PLACEBO

SUMMARY:
Cardiovascular disease (CVD), foremost among which ischemic heart disease and stroke, are the leading cause of mortality and morbidity in France. These diseases are multifactorial origin and even if it is not possible to act on risk markers such as age, sex, or heredity, risk factors like high cholesterol, smoking , hypertension, obesity, diabetes and physical inactivity, are the main target of prevention strategies. Dydlipidemias have a role in the formation of CVD in participating in the genesis of atherosclerosis. The cholesterol and LDL-cholesterol in particular is subject to oxidation process in plasma. The molecules of oxidized LDL-cholesterol, small and dense, easily penetrate the arterial endothelial wall and are greeted by macrophages. Following a succession of different processes including inflammation, atherosclerotic plaque is formed. The result is either an arteriopathy when the arterial lumen narrowing, or atherothrombosis in the event of plaque rupture. Given this pathophysiology, reduce blood lipids, including LDL-cholesterol and reducing oxidation and inflammation are interesting strategies in the context of cardiovascular prevention. Several scientific study showed that nutritional supplementation with some plant extracts such as artichokes, garlic, red yeast rice, or the sugar cane policosanol helps to reduce several cardiovascular risk factors including regulate concentrations of circulating lipids.

In this study, we hypothesize that the food supplement LIMICOL contributes to reducing LDL cholesterol in the context of care for patients (dietary measures and physical activity)

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25 and 35 kg/m²
* Subject has a stable weight for at least three months before the start of the study.
* LDL ≥ 1.50 g/L
* 0.9 g/L ≤ triglycerides ≤ 4.00 g/L
* Subject able and willing to comply with the protocol and agreeing to give his informed consent in writing;
* Subject affiliated with a social security scheme

Exclusion Criteria:

* Subject having a confirmed or suspected food allergy, notably to one of the components of the study product;
* Subject suffering from a severe chronic condition deemed incompatible with participation in the study by the investigator
* Subject with glaucoma
* Subject with uretroprostatic disorder
* Subjet anxious (score >9 HAD scale)
* Subject with diabetes
* Subjet with treatment anticoagulant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
LDL-cholesterol levels (g/l) at the end of study | Week 12
  Effect of LIMICOL supplementation showed by ANCOVA analysis of LDL cholesterol (g/l), with baseline LDL as covariable

SECONDARY OUTCOMES:
Muscle function on tissue biopsy | Week 0; Week 12
  Mitochondrial respiration of muscle histology. Expressed as pmol/s/ml.
Total cholesterol | Week 0; Week 6; Week 12
  Total cholesterol. Expressed as g/l, variation (g/l and %) compared to baseline.
HDL-cholesterol | Week 0; Week 6; Week 12
  HDL. Expressed as g/l, variation (g/l and %) compared to baseline.
Triglycerides | Week 0; Week 6; Week 12
  Triglycerides. Expressed as g/l, variation (g/l and %) compared to baseline.
LDLox | Week 0; Week 6; Week 12
  oxydized LDL. Expressed as pg/ml, variation (pg/l and %) compared to baseline.
CoQ10 | Week 0; Week 12
  circulating coenzyme Q10. Expressed as pg/ml. variation (pg/l and %) compared to baseline.
ApoA1 | Week 0; Week 12
  Circulating ApoLipoprotein A1. Expressed as g/ml. variation (g/l and %) compared to baseline.
ApoB | Week 0; Week 12
  Circulating ApoLipoprotein B. Expressed as g/ml. variation (g/l and %) compared to baseline.
Glycemia | Week 0; Week 12
  Glycemia. Expressed as mmol/l. variation (mmol/l and %) compared to baseline.
Insulinemia | Week 0; Week 12
  Insulinemia. Expressed as mUI/l. variation (mUI/l and %) compared to baseline.
Myoglobin | Week 0; Week 12
  Myoglobin. Expressed as µgI/l. variation (µg/l and %) compared to baseline.
CK | Week 0; Week 12
  Creatin kinase. Expressed as UI/l. variation (UI/l and %) compared to baseline.
LD | Week 0; Week 12
  Lactate Dehydrogenase. Expressed as UI/l. variation (UI/l and %) compared to baseline.
AST | Week 0; Week 12
  Aspartate transaminase. Expressed as UI/l. variation (UI/l and %) compared to baseline.
ALT | Week 0; Week 12
  Alanine transaminase. Expressed as UI/l. variation (UI/l and %) compared to baseline.
ALP | Week 0; Week 12
  Alkaline phosphatase. Expressed as UI/l. variation (UI/l and %) compared to baseline.
GGT | Week 0; Week 12
  Gamma-glutamyltransferase. Expressed as UI/l. variation (UI/l and %) compared to baseline.
Bilirubin | Week 0; Week 12
  Bilirubin. Expressed as µmol/l. variation (µmol/l and %) compared to baseline.
Albumin | Week 0; Week 12
  Albumin. Expressed as g/l. variation (g/l and %) compared to baseline.
Total Protein | Week 0; Week 12
  Total Protein. Expressed as g/l. variation (g/l and %) compared to baseline.
usCRP | Week 0; Week 12
  ultrasensible C-reactiv protein. Expressed as mg/l. variation (mg/l and %) compared to baseline.
Creatinin | Week 0; Week 12
  Creatinin. Expressed as µmol/l. variation (µmol/l and %) compared to baseline.
Urea | Week 0; Week 12
  Urea. Expressed as µmol/l. variation (µmol/l and %) compared to baseline.
VO2 MAX | Week 0; Week 6; Week 12
  VO2MAX. Expressed as ml/min/kg. variation (ml/min/kg and %) compared to baseline.
Max Strength | Week 0; Week 6; Week 12
  Max grip strength. Expressed as N. variation (N and %) compared to baseline.
Weight | Week 0; Week 6; Week 12
  Body Weight. Expressed as Kg. variation (Kg and %) compared to baseline.
Fat mass | Week 0; Week 12
  Fat Mass measured by DEXA. Expressed as % body mass. variation (%) compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Martine Duclos, Pr, Principal Investigator — CHU G. Montpied
Locations (4):
- France (4):
  - Clermont Université, Université Blaise Pascal, EA 3533, Laboratoire des Adaptations Métaboliques à l'Exercice en Conditions Physiologiques et Pathologiques (AME2P), BP 10448, Clermont-Ferrand
  - CRNH-Auvergne, Clermont-Ferrand
  - Service de médecine du sport et des explorations fonctionnelles, CHU G. Montpied, Clermont-Ferrand
  - Clinique de cardiopneumologie de DURTOL, Durtol